CLINICAL TRIAL: NCT01955122
Title: Polyp Detection With the EndoRings™: A Randomized Tandem Colonoscopy Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: EndoAid (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: TSDPR100
Record Dates: First submitted 2013-09-23; First posted 2013-10-07 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2017-03-06 (Actual); Status verified 2017-01

CONDITIONS: Colon Cancer
Keywords: polyp/adenoma miss rate; colonoscopy add-on device; enhanced screening
MeSH Terms: conditions — Colonic Neoplasms; Polyps

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Other): Tandem Colonoscopy- Each patient will undergo 2 colonoscopy procedures:
  a Standard view colonoscopy followed immediately by an EndoRings™ colonoscopy.
  Interventions: Device: Tandem Colonoscopy
- Group B (Other): Tandem Colonoscopy- Each patient will undergo 2 colonoscopy procedures:
  an EndoRings™ colonoscopy followed immediately by a Standard view colonoscopy.
  Interventions: Device: Tandem Colonoscopy

INTERVENTIONS:
Device: Tandem Colonoscopy — Each patient will undergo a double procedure: standard colonoscopy using the EndoRings™ add-on device and Standard colonoscopy (without using the EndoRings™ add-on device) in a randomized order.
  Other Names: Colon screening

SUMMARY:
To compare the adenoma miss rate with the EndoRings™ vs. the adenoma miss rate with Standard view colonoscopy.

To compare the polyp miss rate with the EndoRings™ vs. the polyp miss rate with Standard view colonoscopy.In addition, time measurements including time to cecum, time for withdrawal and overall procedure time will be analyzed and reported for each group.

DETAILED DESCRIPTION:
Patients who are scheduled for screening, surveillance or diagnostic colonoscopy will be recruited to the study and randomized to one of two groups. Each enrolled subject will undergo two "back-to-back" procedures.

Subjects in Group A (study group) will undergo a Standard view colonoscopy followed immediately by an EndoRings™ colonoscopy. Subjects in Group B (control group) will undergo an EndoRings™ colonoscopy followed immediately by a Standard view colonoscopy.

Results from the two groups will be analyzed and compared, with primary outcome measures being adenoma miss rate and polyp miss rate. Secondary outcome measures will include withdrawal time, total procedure time and characteristics of polyps detected, including size and histological results.

Subjects will be followed through a 24 hour and a 7-days telephone interview for analysis of unexpected adverse events. Clinical results will be analyzed using various statistical measures of significance.

Multi-center study with up to 126 patients. Up to 126 treated patients (2 groups of 57 patients +6 drop-out patients) will be enrolled into the study.

ELIGIBILITY:
Inclusion Criteria:

* Subject between the ages of 40 and 75
* The patient is undergoing colonoscopy for screening, for surveillance in follow-up of previous polypectomy or for diagnostic workup;
* Written informed consent must be available before enrollment in the trial

Exclusion Criteria:

* Patients with a history of colonic resection;
* Patients with known (or newly diagnosed) inflammatory bowel disease;
* Patients with a personal history of polyposis syndrome;
* Patients with suspected chronic stricture potentially precluding complete colonoscopy;
* Patients with diverticulitis or toxic megacolon;
* Patients with a history of radiation therapy to abdomen or pelvis;
* Patients with a hemorrhagic diathesis
* Patients with acute lower GI bleeding
* Pregnant women and women with childbearing potential without adequate contraception
* Patients who are currently enrolled in another clinical investigation in which the intervention might compromise the safety of the patient's participation in this study.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Meytal Segev, DMD, Study Director — EndoAid Ltd.; Ian Gralnek, Prof., Principal Investigator — Rambam Health Care Campus; Ori Segol, Dr., Principal Investigator — Carmel Medical Center; Peter Siersema, Prof., Principal Investigator — UMC Utrecht; Douglas K. Rex, Dr., Principal Investigator — Indiana University
Locations (3):
- Indiana University, Indianapolis, Indiana, United States
- Elisha Medical Center, Haifa, Please Select, Israel
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dik VK, Gralnek IM, Segol O, Suissa A, Belderbos TD, Moons LM, Segev M, Domanov S, Rex DK, Siersema PD. Multicenter, randomized, tandem evaluation of EndoRings colonoscopy--results of the CLEVER study. Endoscopy. 2015 Dec;47(12):1151-8. doi: 10.1055/s-0034-1392421. Epub 2015 Jul 28. PMID 26220283

RESULTS

PARTICIPANT FLOW:
Groups:
- Group B: Tandem Colonoscopy: Each patient will undergo 2 colonoscopy procedures:
  an EndoRings™ colonoscopy followed immediately by a Standard view colonoscopy.
Period: Overall Study
Arm/Group | Group A | Group B
Started | 64 (Excluded (n = 5) Included in analysis (n = 59)) | 62 (Excluded (n = 5) Included in analysis (n = 57))
No.Patients Enrolled | 64 | 62
No. Patients Completed Double Procedure | 59 | 57
Completed | 59 | 57
Not Completed | 5 | 5
Not completed — Physician Decision | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Group A: Tandem Colonoscopy: Each patient will undergo a double procedure: Standard colonoscopy (without using the EndoRings™ add-on device) followed by EndoRings™ colonoscopy.
- Group B: Tandem Colonoscopy: Each patient will undergo a double procedure: EndoRings™ colonoscopy followed by Standard colonoscopy (without using the EndoRings™ add-on device) .
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 59 | 57 | 116
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 40 | 80
  >=65 years | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (9.3) | 57.9 (9.1) | 58.7 (9.2)
Gender [Count of Participants; unit: Participants]
  Female | 29 | 16 | 45
  Male | 30 | 41 | 71
Region of Enrollment [Number; unit: participants]
  Netherlands | 34 | 36 | 70
  United States | 5 | 3 | 8
  Israel | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Adenoma and Polyp Miss Rate
Description: Group A- we measured the Adenoma&Polyp miss rates in the first procedure with Standard (based on what we discovered on the second procedure with the EndoRings).
  Group B- we measured the Adenoma&Polyp miss rates in the first procedure with EndoRings (based on what we discovered on the second procedure with the Standard).
  Adenoma/Polyp Miss Rate means: total number of adenomas or polyps detected during the second procedure per Group divided by the total number of adenomas/polyps detected overall per Group]*100
Time Frame: 30min for Standard colonoscopy and 30min for EndoRings colonoscopy- 1 hour in total.
Measure: Number (95% Confidence Interval); unit: percentage of :Adenomas/Polyp missed
Arm/Group | Group A | Group B
Number analyzed (Participants) | 59 | 57
percentage of :Adenomas/Polyp missed
  Adenoma Miss Rate | 48.3 [35.0 to 61.2] | 10.4 [2.9 to 18.0]
  Polyp Miss Rate | 52.8 [43.2 to 62] | 9.1 [3.9 to 14.3]

2. Secondary Outcome: Total Number of Therapeutic Interventions Performed
Description: Ability to perform therapeutic interventions, such as biopsies, polypectomies, APC etc. during the Standard Colonoscopy and during the EndoRings Colonoscopy. The number of interventions was not compared, this was just a safety outcome meant to prove there was no difficulty in performing interventions in both arms.
Time Frame: Interventions during procedure
Measure: Number; unit: Total Interventions performed
Arm/Group | Group A | Group B
Number analyzed (Participants) | 59 | 57
Total Interventions performed | 106 | 121

3. Secondary Outcome: Procedure Time A Stopwatch Will be Used for Stopping the Timing of the Procedure for Any Polypectomy Performed and Then Restarting Once the Polypectomy is Completed, Meaning That Purely Procedure Time is Measured
Description: The following will be recorded: a. Time for intubation to the cecum. b. Time for withdrawal from the cecum to the anal verge. c. Total procedure time A stopwatch will be used for stopping the timing of the procedure for any polypectomy performed and then restarting once the polypectomy is completed, meaning that purely procedure time is measured
Time Frame: During the procedure
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- EndoRings Colonoscopy: procedures performed with the EndoRings
- Standard Colonoscopy: procedures performed with the Standard
Arm/Group | EndoRings Colonoscopy | Standard Colonoscopy
Number analyzed (Participants) | 116 | 116
minutes
  Total procedure time | 21.6 (8.9) | 18.5 (8.2)
  Time to cecum | 9.3 (7.3) | 8.4 (5.6)
  Withdrawal time | 7.4 (1.9) | 7.2 (2.2)

4. Secondary Outcome: Sedation
Description: Sedation dosage
Time Frame: During the procedure
Population: Sedation dosage was not collected from any participant during the study
Groups:
- Group B: Tandem Colonoscopy: Each patient will undergo a double procedure: EndoRings™ colonoscopy followed by Standard colonoscopy (without using the EndoRings™ add-on device).
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Scope Centering Ability
Description: Ability to center the scope inside the gastrointestinal tract.
Time Frame: During the procedure
Population: Centering ability was not collected from any procedure during the study
Groups:
- Group A: Tandem Colonoscopy- Each patient will undergo 2 colonoscopy procedures:
  a Standard view colonoscopy followed immediately by an EndoRings™ colonoscopy.
  Tandem Colonoscopy: Each patient will undergo a double procedure: standard colonoscopy using the EndoRings™ add-on device and Standard colonoscopy (without using the EndoRings™ add-on device) in a randomized order.
- Group B: Tandem Colonoscopy- Each patient will undergo 2 colonoscopy procedures:
  an EndoRings™ colonoscopy followed immediately by a Standard view colonoscopy.
  Tandem Colonoscopy: Each patient will undergo a double procedure: standard colonoscopy using the EndoRings™ add-on device and Standard colonoscopy (without using the EndoRings™ add-on device) in a randomized order.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Colon Area Screened
Description: Subjective evaluation of the additional area screened by the physician.
Time Frame: During the procedure
Population: Evaluation of the additional area screened by the physician was not collected from any participant during the study
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Patient Satisfaction
Description: Follow up phone call was done 24 hours post procedure. Patients were asked the following : "On a 0 to 10 scale, with "0" being no pain and "10" being pain as bad as you can imagine, how would you describe your colonoscopy experience?" 0 1 2 3 4 5 6 7 8 9 10
Time Frame: 24 hours post procedure
Population: Data was not analyzed since the patients satisfactory score was general estimation which could not be associated with either the standard colonoscopy or the EndoRings colonoscopy, therefore the intended endpoint failed.
Arm/Group | Group A | Group B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 hours post procedure
Description: Serious or Other (non-serious) Adverse Events were monitored/assessed, but none were observed
Groups:
- A (Study Group): Tandem Colonoscopy: Each patient will undergo a double procedure: Standard colonoscopy (without using the EndoRings™ add-on device) followed by EndoRings™ colonoscopy.
- Group B (Control Group): Tandem Colonoscopy: Each patient will undergo a double procedure: EndoRings™ colonoscopy followed by Standard colonoscopy (without using the EndoRings™ add-on device).
Arm/Group | A (Study Group) | Group B (Control Group)
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/57
Other Adverse Events (participants affected / at risk) | 0/59 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days